CLINICAL TRIAL: NCT05216133
Title: AERODIGESTIVE DISEASE IN THE WORLD TRADE CENTER EXPOSED FDNY COHORT: a Single Center Observational Study of Biomarkers of Airway Disease, Barrett's and Underdiagnosed Reflux Noninvasively (BADBURN)
Brief Title: Biomarkers of Airway Disease, Barrett's and Underdiagnosed Reflux Noninvasively (BADBURN)
Status: Enrolling by invitation | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 21-00679
Record Dates: First submitted 2022-01-18; First posted 2022-01-31 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Airway Disease; Barrett Esophagus; Gastroesophageal Reflux Disease
MeSH Terms: conditions — Barrett Esophagus; Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, salivary samples, exhaled breath condensate (EBC), nasopharyngeal and oropharyngeal swabs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A majority of Fire Department of New York (FDNY) World Trade Center (WTC) exposed rescue and recovery workers developed gastroesophageal reflux disease (GERD), a risk factor for Barrett's Esophagus (BE) and subsequent esophageal cancer. There is diminished health-related quality of life and productivity associated with aerodigestive diseases such as GERD and BE.

This proposal will leverage the longitudinally phenotyped WTC exposed cohort, validate biomarkers of WTC-aerodigestive disease, and develop novel, noninvasive disease phenotyping of premalignant diseases such as BE, and identify potential targeted therapeutics to improve care.

ELIGIBILITY:
Inclusion Criteria:

1. Age 37-90
2. FDNY rescue and recovery worker.
3. Male*
4. Documented WTC exposure.
5. Consented/Enrolled in the FDNY WTC Health Program
6. Subjects are willing and able to consent for themselves to study enrollment
7. Subjects are willing and able to participate in study procedures
8. Are able to perform their activities of daily living independently
9. Are either light duty or retired FDNY Firefighters
10. Spirometry available within the last 24 months, and at a post-9/11 visit.
11. Have means to accommodate transportation to/from in-person visit Are able to attend a single visit at the CTSI (462 1st Avenue, C & D 4th Floor)
12. Pre-9/11 spirometry with FEV1%predicted ≥LLN and if not available 1st -post 9/11 spirometry with an FEV1 >80% predicted.
13. Exposure at the WTC-site within 2 weeks of the 9/11/2001
14. Entered WTC-HP before the site closure on 7/24/2002.
15. Serum from their first post 9/11 WTC-HP visit is available in the FDNY WTC biorepository and may be assayed
16. Are not currently being treated for malignancy
17. Subjects will either need to be defined as having WTC-AHR, WTC-GERD, WTC-BE or be designated controls as per the following additional inclusion criteria are specific to the WTC-aerodigestive disease that the subjects have
18. AHR--A positive methacholine (PC20<16) and/or positive bronchodilator response (ATS/ERS guidelines: improvement of FEV1 by 12% and at least 200mL) at least once post-9/11.[95, 96]No recorded positive AHR testing prior to 9/11
19. GERD Inclusion Criteria

    * Erosive esophagitis LA grade C or D (as described on endoscopy), OR
    * Stricture or Barrett's esophagus on endoscopy, OR
    * Esophageal acid exposure time >6% on a pH or pH impedance study

19. BE Inclusion Criteria

* Columnar epithelium lining ≥1 cm of the distal esophagus. AND
* Histologic examination of biopsy specimens from that columnar epithelium must reveal intestinal metaplasia characterized with goblet cells.

Exclusion Criteria:

1. Unwilling to complete an informed consent.
2. Not enrolled in the WTC-HP
3. Do not meet eligibility criteria for AIM 1 or did not have serum available in the biorepository from the first post 9/11 WTC-HP visit.
4. Have pre-existing and documented conditions or concurrent diagnoses, including (and not necessarily limited to) active cancer, severe heart disease, significant cognitive impairment, eating disorders, significant psychiatric illness, end-stage COPD, severe pulmonary hypertension, or organ transplant.
5. High dose steroid (>20mg prednisone or equivalent) or other hormonal treatments/chemotherapy use in the last month, including testosterone supplementation.
6. Life-expectancy < 6 months
7. Female*

Ages: 37 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Less than 1 % of the FDNY-HP subjects are female. As such our prior work has excluded females. In addition, due to this small sample size and since there is significant literature that biomarkers are different in these two sexes, the study team will not be enrolling females.
Study Population: Male FDNY rescue and recovery workers between the ages of 37 and 90.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-03-22 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Levels of salivary pepsin | up to Day 365
  Saliva will be analyzed using the Peptest. The value of >/= 16 ng/mL indicates a positive salivary pepsin.
pH Levels from Exhaled Breath Condensate (EBC) | up to Day 365
  EBC pH assay will be performed
Histamine Concentration from Exhaled Breath Condensate (EBC) | up to Day 365
  Histamine concentration will be measured with an enzymatic immunoassay
Score on Patient Assessment of Upper Gastrointestinal Disorders-Quality of Life (PAGI-QOL) Questionnaire | up to Day 365
  PAGI-QOL asks about how some of the gastrointestinal problems one may be experiencing (such as pain, discomfort, or other problems) may have affected one's overall quality of life and well-being in the past 2 weeks. PAGI-QOL consists of 30 questions, each scored from 0 (none of the time) to 5 (all of the time). The total score range is 0-150; the higher the score, the less the quality of life and well-being.
Score on Patient Assessment of Upper Gastrointestinal Disorders-Symptoms (PAGI-SYM) Questionnaire | up to Day 365
  PAGI-SYM asks about the severity of symptoms one may have related one's gastrointestinal problem. The questionnaire consists of 20 symptoms, and each symptom is scored from 0 (none) to 5 (very severe). The total score range is 0-100; the higher the score, the more severe the symptoms.
Score on St. George's Respiratory Questionnaire (SGRQ-C) | up to Day 365
  SGRQ-C is designed to assess how one's breathing is troubling a participant and how it affects one's life. The questionnaire consists of 14 questions. The total score range is 0-54; the higher the score, the worse the chest trouble.
36-Item Short Form Survey Instrument (SF-36) | up to Day 365
  SF-36 captures mental health, general health perception, emotional, and social role functioning. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Nolan, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Clinical & Translational Science Institute Clinical Research Center (CTSI CRC), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose will have access to the data to achieve aims in the approved proposal. Requests should be directed to anna.nolan@med.nyu.edu. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Javed U, Podury S, Kwon S, Liu M, Kim DH, Fallahzadeh A, Li Y, Khan AR, Francois F, Schwartz T, Zeig-Owens R, Grunig G, Veerappan A, Zhou J, Crowley G, Prezant DJ, Nolan A. Biomarkers of Airway Disease, Barrett's and Underdiagnosed Reflux Noninvasively (BAD-BURN) in World Trade Center exposed firefighters: a case-control observational study protocol. BMC Gastroenterol. 2024 Aug 9;24(1):255. doi: 10.1186/s12876-024-03294-9. PMID 39123126
- [Derived] Javed U, Podury S, Kwon S, Liu M, Kim D, Fallah Zadeh A, Li Y, Khan A, Francois F, Schwartz T, Zeig-Owens R, Grunig G, Veerappan A, Zhou J, Crowley G, Prezant D, Nolan A. Biomarkers of Airway Disease, Barrett's and Underdiagnosed Reflux Noninvasively (BAD-BURN): a Case-Control Observational Study Protocol. Res Sq [Preprint]. 2024 May 15:rs.3.rs-4355584. doi: 10.21203/rs.3.rs-4355584/v1. PMID 38798396